CLINICAL TRIAL: NCT03523351
Title: A Randomized Trial of Early, Upfront Palliative Radiation Therapy Versus Standard of Care for Patients With Highest Risk Asymptomatic or Minimally Symptomatic Bone Metastases
Brief Title: Study of Palliative Radiation Therapy vs. no Palliative Radiation Therapy for Patients With High Risk Bone Metastases That Are Not Causing Significant Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-196
Record Dates: First submitted 2018-05-01; First posted 2018-05-14 (Actual); Results first posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Solid Tumors of Metastatic Disease
Keywords: Palliative Radiation; 18-196
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: In this trial patients will be divided into 2 cohorts. Patients in Cohort 1 will undergo standard of care therapy for bone metastases. Patients in Cohort 2 will undergo upfront RT to ≤5 highest risk bone metastases first followed by standard of care therapy.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of care (Active Comparator): Patients randomized to Arm 1 will undergo appropriate therapy as determined by their oncologist. These patients will either continue their current therapy or be transitioned to a new standard of care therapy at the discretion of the treating oncologist. If randomized to Arm 1, these patients may undergo palliative RT for progressive, painful lesions (a skeletal related event) at time of symptom development (not upfront palliative RT).
  Interventions: Drug: Systemic Therapy
- Selective radiation to ≤5 highest risk bone metastases (Experimental): Patients on Arm 2 of the study will undergo selective RT to ≤ 5 high risk bone metastases defined as 1. bulkiest sites of osseous disease ≥ 2cm, 2. disease involving the hip (acetabulum, femoral head, femoral neck), shoulder (acromion, glenoid, humeral head), or sacroiliac joints 3. disease in long bones with1/3-2/3 cortical thickness (humerus, radius, ulna, clavicle, femur, tibia, fibula, metacarpus, phalanges) 4. disease in junctional spine (C7-T1, T12-L1, L5-S1) &/or disease with posterior element involvement.
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — Radiation therapy will be delivered according to department standards. For this protocol, total dose and dose fractionation may be delivered at the discretion of the treating radiation oncologist according to department standards. All techniques including conventional, 3D-CRT, or IMRT technique may be used. Image guidance at the time of treatment delivery to verify patient positioning may be chosen at the discretion of the treating radiation oncologist according to department standards.
  Arms: Selective radiation to ≤5 highest risk bone metastases
Drug: Systemic Therapy — Standard of care systemic therapy, including chemotherapeutics, targeted therapies, immunomodulatory agents, and hormonal therapies will be delivered at the discretion of the treating medical oncologist. Patients may receive systemic therapy concurrently and there are no restrictions on initiation of systemic agents after radiotherapy including immunotherapy and hormonal therapy, the timing of which will be determined by a consensus between the treating medical and radiation oncologists.
  Arms: Standard of care

SUMMARY:
The purpose of the study is to compare the outcome of patients who receive standard treatment versus those who receive preventative radiation and then standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor malignancy with greater than 5 sites of metastatic disease detected on imaging.
* Has high risk bone metastases that are asymptomatic or minimally symptomatic (not requiring opioids). High risks metastases are defined as: 1. bulkiest sites of osseous disease ≥ 2cm, 2. disease involving the hip (acetabulum, femoral head, femoral neck), shoulder (acromion, glenoid, humeral head), or sacroiliac joints 3. disease in long bones with1/3-2/3 cortical thickness (humerus, radius, ulna, clavicle, femur, tibia, fibula, metacarpus, phalanges) 4. disease in junctional spine (C7-T1, T12-L1, L5-S1) and/or disease with posterior element involvement.
* ECOG performance status 0 - 2.
* Age ≥ 18 years.
* Able to provide informed consent.
* Patients at reproductive potential must agree to practice an effective contraceptive method. Women of childbearing potential must not be pregnant or lactating.

Exclusion Criteria:

* Previous radiotherapy to the intended treatment site that precludes developing a treatment plan that respects normal tissue tolerances.
* Serious medical co-morbidities precluding radiotherapy.
* Pregnant or lactating women.
* Target lesion(s) is/are complicated bone metastases that include clinical or radiological evidence of spinal cord compression or impending pathological fracture.
* Leptomeningeal disease.
* Malignant pleural effusion.
* Absolute neutrophil count (ANC) <1.0 K/mcL and platelet count <50 K/mcL at time of enrollment.
* Patients whose entry to the trial will cause unacceptable clinical delays in their planned management.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Divya Yerramilli, MD, MBE, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - Baptist Alliance Miami Cancer Institute, Miami, Florida
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Lehigh Valley Health Network, Allentown, Pennsylvania

REFERENCES:
- [Derived] Gillespie EF, Yang JC, Mathis NJ, Marine CB, White C, Zhang Z, Barker CA, Kotecha R, McIntosh A, Vaynrub M, Bartelstein MK, Mitchell A, Guttmann DM, Yerramilli D, Higginson DS, Yamada YJ, Kohutek ZA, Powell SN, Tsai J, Yang JT. Prophylactic Radiation Therapy Versus Standard of Care for Patients With High-Risk Asymptomatic Bone Metastases: A Multicenter, Randomized Phase II Clinical Trial. J Clin Oncol. 2024 Jan 1;42(1):38-46. doi: 10.1200/JCO.23.00753. Epub 2023 Sep 25. PMID 37748124
- [Derived] Rosen DB, Benjamin CD, Yang JC, Doyle C, Zhang Z, Barker CA, Vaynrub M, Yang TJ, Gillespie EF. Early palliative radiation versus observation for high-risk asymptomatic or minimally symptomatic bone metastases: study protocol for a randomized controlled trial. BMC Cancer. 2020 Nov 17;20(1):1115. doi: 10.1186/s12885-020-07591-w. PMID 33203426
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care | Selective Radiation to ≤5 Highest Risk Bone Metastases
Started | 39 | 39
Completed | 20 | 23
Not Completed | 19 | 16
Not completed — Death | 13 | 11
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Patient was not treated on study but enrolled due to progressive disease during active treatment | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Selective Radiation to ≤5 Highest Risk Bone Metastases | Total
Number analyzed (Participants) | 39 | 39 | 78
Age, Continuous [Mean (Full Range); unit: years] | 58 [37 to 78] | 58 [38 to 84] | 58 [37 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 22 | 21 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 8
  Not Hispanic or Latino | 33 | 35 | 68
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 6 | 10
  White | 32 | 28 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39 | 39 | 78

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Skeletal Related Events (SREs)
Description: which will be defined as pathological fractures, spinal cord compression, or palliative radiotherapy and orthopedic surgery to bone.
Time Frame: 1 year
Measure: Number; unit: number of participants
Arm/Group | Standard of Care | Selective Radiation to ≤5 Highest Risk Bone Metastases
Number analyzed (Participants) | 39 | 39
number of participants
  Skeletal Related Events | 10 | 1
  No Skeletal Related Events | 29 | 38

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Standard of Care | Selective Radiation to ≤5 Highest Risk Bone Metastases
All-Cause Mortality (participants affected / at risk) | 28/39 | 19/39
Serious Adverse Events (participants affected / at risk) | 4/39 | 2/39
Other Adverse Events (participants affected / at risk) | 34/39 | 35/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (N=39) | Selective Radiation to ≤5 Highest Risk Bone Metastases (N=39)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Esophageal varices (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Esophagitis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Neutrophil count decrease (Investigations) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (N=39) | Selective Radiation to ≤5 Highest Risk Bone Metastases (N=39)
Anemia (Blood and lymphatic system disorders) | 28 | 26
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Buttock Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 4 | 8
Fatigue (General disorders) | 11 | 22
Hyponatremia (Metabolism and nutrition disorders) | 9 | 7
Lymphocyte count decreased (Investigations) | 22 | 24
Nausea (Gastrointestinal disorders) | 3 | 7
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 5 | 6
Pain (General disorders) | 5 | 6
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 1
Platelet count decreased (Investigations) | 10 | 10
Vomiting (Gastrointestinal disorders) | 1 | 2
White blood cell decreased (Investigations) | 12 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-05): https://cdn.clinicaltrials.gov/large-docs/51/NCT03523351/Prot_SAP_000.pdf